CLINICAL TRIAL: NCT01519752
Title: A Randomized, Double-Blind, Placebo Controlled, Parallel Design, Multiple-Site, Study Comparing Oxiconazole Nitrate Cream 1% (Taro Pharmaceuticals,Inc) to Oxistat® (Oxiconazole Nitrate Cream) Cream 1% (PharmaDerma) in the Treatment of Tinea Pedis
Brief Title: A Therapeutic Equivalence Study of Two Oxiconazole Nitrate Topical Cream Treatments for Patients With Tinea Pedis
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: OXZC 1102
Record Dates: First submitted 2012-01-19; First posted 2012-01-27 (Estimated); Last update posted 2014-01-22 (Estimated); Status verified 2014-01

CONDITIONS: Tinea Pedis
Keywords: Tinea Pedis
MeSH Terms: conditions — Tinea Pedis | interventions — oxiconazole

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Oxiconazole Nitrate Cream 1% (Experimental)
  Interventions: Drug: Oxiconazole Nitrate Cream 1%
- Oxiconazole Nitrate Cream 1% (Oxistat®) (Active Comparator)
  Interventions: Drug: Oxiconazole Nitrate Cream 1% (Oxistat®)
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxiconazole Nitrate Cream 1% — Oxiconazole Nitrate Cream 1% applied to affected area once a day for 28 days
  Arms: Oxiconazole Nitrate Cream 1%
Drug: Oxiconazole Nitrate Cream 1% (Oxistat®) — Oxiconazole Nitrate Cream 1%(Oxistat®)applied to affected area once a day for 28 days
  Arms: Oxiconazole Nitrate Cream 1% (Oxistat®)
Drug: Placebo — Placebo applied to affected area once a day for 28 days
  Arms: Placebo

SUMMARY:
The objective of this study is to demonstrate that Oxiconazole nitrate 1% topical cream is effective for the treatment of patients with moderate to severe Tinea pedis.

ELIGIBILITY:
Inclusion Criteria:

1. Male or non-pregnant, non-lactating female, 12 years of age or older.
2. Signed informed consent form, which meets all criteria of current FDA regulations
3. If female and of child bearing potential, prepare to abstain from sexual intercourse or use a reliable method of contraception during the study {e.g., condom, IUD, oral, transdermal, injected or implanted hormonal contraceptives)and (must have used the same product for at least 30 days prior to the study start and use the same product throughout the duration of the study), transdermal or implanted hormonal contraceptives}
4. A confirmed clinical diagnosis of tinea pedis with lesions localized to the interdigital spaces or predominantly interdigital, but may extend to other areas of the foot. (the non-interdigital lesions should not be hyperkeratotic i.e., characteristic of moccasin).
5. The presence of tinea pedis infection, confirm by the observation of segmented fungal hyphae during a microscopic KOH wet mount examination.

Exclusion Criteria:

1. Females who are pregnant, or lactating or likely to become pregnant during the study.
2. Any known hypersensitivity to oxiconazole nitrate or other antifungal agents.
3. Patients with a past history of tinea pedis infections with a lack of response to antifungal therapy (i.e. recurrent tinea pedis, more than 3 infections in the past 12 months, which were unresponsive to previous antifungal therapy).
4. Participation in a research study in the past 30 days prior to screening/randomization.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 661 (Actual)
Dates: Start 2011-11; Primary Completion 2012-08 (Actual); Study Completion 2012-11 (Actual)

PRIMARY OUTCOMES:
Therapeutic Cure | Day 42
  Clinical & Mycological Cure at 6 weeks

SECONDARY OUTCOMES:
Clinical Cure | Day 42
  Proportion of patients considered a clinical cure at 6 weeks
Mycological Cure | Day 42
  Proportion of patients with both KOH & culture negative at 6 weeks